CLINICAL TRIAL: NCT01985555
Title: A Phase I, Open-label, Multicenter Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of Volitinib in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of the Volitinib (HMPL-504) in Patients With Advanced Solid Tumors
Acronym: HMPL-504
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-504-00CH1
Record Dates: First submitted 2013-11-01; First posted 2013-11-15 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-02

CONDITIONS: Tumors
Keywords: Phase I; Safety; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volitinib(HMPL-504) (Experimental): There are 5 dose cohorts,including600 QD,800QD and 400BID mg,500BID in the dose escalation stage and HMPL-504 will be administered orally to patients once daily for each dose cohort., in the dose expansion stage 500BID will be administered orally to patients.
  Interventions: Drug: Volitinib(HMPL-504)

INTERVENTIONS:
Drug: Volitinib(HMPL-504) — Volitinib(HMPL-504) is a tablet in the form of 25 mg ,100mg and 200 mg,oral,once daily or 2 times a day.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple doses of volitinib administered to patients with locally advanced or metastatic solid tumors and determine MTD (Maximum Tolerated Dose) or RPTD(recommended Phase 2 dose).

DETAILED DESCRIPTION:
The primary endpoint is evaluation of safety and tolerability during all the study of therapy following the initiation of multiple dosing of HMPL-504. The safety and tolerability variables to be evaluated in this study are adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology (Maximum Tolerated Dose), and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for protein), and electrocardiograms (ECGs) in triplicate, Incidence and nature of DLTs (Dose-Limiting Toxicity), to determine the MTD (Maximum Tolerated Dose).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age≥18 years
* Histologically or cytologically documented(include both dose escalation stage and dose expansion stage), incurable, locally advanced, or metastatic solid malignancy
* In the dose escalation stage: patients with any malignant solid tumor type for whom standard therapy either has proven to be ineffective (progressed on, or failed to respond to) or intolerable, have no access to standard systemic therapy or standard systemic therapy does not exist.
* In the dose expansion stage:

Metastatic or locally advanced gastric cancer patients with cMet positive b)Metastatic or locally advanced EGFR wild type NSCLC patients and with cMet positive.

* ECOG performance status of 0, or 1
* Male or female patients of child-producing potential must agree to use double barrier contraception, condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD), contraceptives (oral or parenteral), Implanon, injectables or other avoidance of pregnancy measures during the study and for 90 days after the last day of treatment

Exclusion Criteria:

* Absolute neutrophil count <1500 cells/uL, hemoglobin <9 g/dL or platelet count < 100,000/mm3
* Total bilirubin > 1.5×the the upper limit of normal(ULN).
* Herbal therapy <1 week prior to Day 1
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia
* Clinical significant active infection
* Known clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus infection
* Pregnant (positive pregnancy test) or lactating women
* Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Involved in other clinical trials < 4weeks prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is evaluation of safety and tolerability during all the study of therapy following the initiation of multiple dosing of Volitinib (HMPL-504). | up to 20 months
  The primary endpoint is evaluation of safety and tolerability during all the study of therapy following the initiation of multiple dosing of HMPL-504. The safety and tolerability variables to be evaluated in this study are adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology(Maximum Tolerated Dose) , and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for protein), and electrocardiograms (ECGs) in triplicate,Incidence and nature of DLTs(Dose-Limiting Toxicity),To determine the MTD (Maximum Tolerated Dose).

SECONDARY OUTCOMES:
Pharmacokinetic Assessments for area under curve (AUC), Cmax and Tmax . | Day 1-3 Single Dose and Day 1-21 Steady State
  In the study of single-dose, full Pharmacokinetics(PK) profiles of HMPL-504 will be obtained following administration of a single oral dose of HMPL-504 on Day 1 to Day 3. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5,2,4,6,8 hour time points on days 1,15,21of dosing in the first 21-Day cycle of therapy, and pre-dose on days 2,8,16,and 22 of the first 21-Day cycle of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD.PHD, Principal Investigator — Investigator
Locations (1):
- BeijingCancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No